CLINICAL TRIAL: NCT02739685
Title: Everolimus-eluting Bioresorbable Vascular Scaffolds Versus Everolimus-eluting Stents in Patients With Chronic Total Occlusion
Brief Title: Bioresorbable Vascular Scaffolds Versus Stents in Patients With Chronic Total Occlusion
Acronym: SCORE-CTO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment, access to devices
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Holger Thiele, Director, Department of Cardiology/Angiology/Intensive Care Medicine, University Heart Center Luebeck, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-373
Record Dates: First submitted 2016-04-13; First posted 2016-04-15 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bioresorbable vascular scaffold (Experimental): Implantation of everolimus-eluting bioresorbable vascular scaffold in chronic total occlusion
  Interventions: Device: Everolimus-eluting bioresorbable vascular scaffold
- Stent (Active Comparator): Implantation everolimus-eluting stent in chronic total occlusion
  Interventions: Device: Everolimus-eluting stent

INTERVENTIONS:
Device: Everolimus-eluting bioresorbable vascular scaffold — Implantation of everolimus-eluting bioresorbable vascular scaffold in chronic total occlusion
  Arms: Bioresorbable vascular scaffold
Device: Everolimus-eluting stent — Implantation of everolimus-eluting stent in chronic total occlusion
  Arms: Stent

SUMMARY:
The purpose of the current study is to demonstrate non-inferiority of everolimus-eluting bioresorbable vascular scaffold to everolimus-eluting stents in patients with chronic total occlusion regarding the antirestenotic efficacy at 8 to 10-month angiographic follow-up.

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria:

* Age ≥18 years
* Angina pectoris, equivalent symptoms, and/or positive stress test
* Viable myocardium subtended by chronic total occlusion
* Negative pregnancy test in women with childbearing potential

Angiographic inclusion criteria:

* Chronic total occlusion defined as Thrombolysis in Myocardial Infarction flow 0 with an estimated duration ≥3 months
* Successful wire passage and assumption of successful stent/scaffold deployment
* Target reference vessel diameter 2.5 - 4.0 mm

Exclusion Criteria:

Clinical exclusion criteria:

* Limited long-term prognosis with a life-expectancy <12 months
* Contraindications to antiplatelet therapy
* Known allergy against cobalt chrome, everolimus, or polylactic acid

Angiographic exclusion criteria:

* Target lesion located in the left main trunk
* Target lesion located in a coronary bypass graft
* Bifurcation lesion with planned two-stent strategy
* Indication for coronary artery bypass grafting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
In-stent late lumen loss assessed by angiography | 8-10 months after the index procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Luebeck, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: Undecided